CLINICAL TRIAL: NCT04531644
Title: Impact of Double Stimulation (DuoStim) in Women Affected by Low Prognosis to Assisted Reproductive Technologies
Brief Title: Double Stimulation in Women With Low Prognosis in ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tu Du Hospital (Other Government)
Collaborators: Federico II University (Other); University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Thi Minh Chau, Head of department of Infertility, Tu Du Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/TD/20/05
Record Dates: First submitted 2020-08-18; First posted 2020-08-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Assisted Reproductive Techniques
Keywords: double ovarian stimulation; low prognosis women; ongoing pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): the patients in this group will be treated with double stimulation
  Interventions: Procedure: double stimulation
- Control (Active Comparator): the patients in this group will be treated with conventional ovarian stimulation
  Interventions: Procedure: conventional ovarian stimulation

INTERVENTIONS:
Procedure: double stimulation — the patients will be treated with two consecutive ovarian stimulations in one cycle
  Other Names: DuoStim
  Arms: Study
Procedure: conventional ovarian stimulation — the patients will be treated with one conventional ovarian stimulation in one cycle
  Arms: Control

SUMMARY:
The main objective of this study is to compare the cumulative ongoing pregnancy rates of two different IVF protocols in women candidate for ART characterized by low prognosis.

DETAILED DESCRIPTION:
The patients will be allocated into two groups: control and study group _ In study group, patients will be treated by DuoStim protocol: The first phase of ovarian stimulation is started on the second day or third day of period. GnRH agonist will be used to trigger when at least two follicles ≥ 17 mm. Approximately 36 hours later, oocytes will be retrieved vaginally under ultrasound monitoring and ICSI will be performed. Five days later after oocyte retrieval, the second stimulation will be started. All embryos will be cryopreserved.

_ In control group, patients will be treated with antagonist protocol: The cycle of ovarian stimulation is started on the second day or third day of period. hCG will be used to trigger when at least two follicles ≥ 17 mm. Approximately 36 hours later, oocytes will be retrieved vaginally under ultrasound monitoring and ICSI will be performed. If serum progesterone on the day of trigger ≥ 1.5 ng/ml, all embryos will be cryostored; otherwise, fresh embryos will be transferred.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 40.
* AMH ≥ 0.3 ng/ml and ≤ 1.2 ng/ml.
* OR 3 ≤ AFC ≤7.
* Normal shape of uterus (based on ultrasound).
* Body mass index within 28 - 37 kg/m2

Exclusion Criteria:

* Asherman's syndrome.
* Endometriosis.
* Leiomyomas distorting the endometrium
* Sperm extracted from surgical procedures (i.e. PESA, TESE).
* Patients refuse to continue participating in the study.
* Patients injected with wrong dose of gonadotropins during the treatment.
* Serious complications or accidents arise forcing the patients to discontinue the treatments.
* Ovarian surgery
* Previous chemotherapy or pelvic irradiation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative Ongoing pregnancy rate | week 11 - 14 of pregnancy
  calculated by the number of ongoing pregnancy patients divided by the total number of patients in appropriate group

SECONDARY OUTCOMES:
Pregnancy rate | 2 weeks after embryo transfer
  beta-hCG test is positive
Ongoing pregnancy rate | week 11 - 14 of pregnancy
  defined as the pregnancy completed 11 - 14 weeks of gestation and having vital fetus
Number of oocytes retrieved | 4 hours after occyte pick-up
  Number of oocytes retrieved identified by the embryologists
Number of mature oocytes | 4 hours after oocyte pick-up
  Number of mature oocytes identified by the embryologists
Number of competent embryos | 3 days to 5 days after oocyte pick-up
  Number of embryos that can be transferred
Fertilization rate | 1 to 3 days after oocyte pick-up
  number of fertilized oocyted divided by number of mature oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Chau TM Le, PhD, Study Director — Tu Du Hospital
Locations (1):
- Department of Infertility of Tu Du hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cardoso MCA, Evangelista A, Sartorio C, Vaz G, Werneck CLV, Guimaraes FM, Sa PG, Erthal MC. Can ovarian double-stimulation in the same menstrual cycle improve IVF outcomes? JBRA Assist Reprod. 2017 Sep 1;21(3):217-221. doi: 10.5935/1518-0557.20170042. PMID 28837031
- [Result] Kuang Y, Chen Q, Hong Q, Lyu Q, Ai A, Fu Y, Shoham Z. Double stimulations during the follicular and luteal phases of poor responders in IVF/ICSI programmes (Shanghai protocol). Reprod Biomed Online. 2014 Dec;29(6):684-91. doi: 10.1016/j.rbmo.2014.08.009. Epub 2014 Sep 6. PMID 25444501
- [Result] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Result] Ubaldi FM, Capalbo A, Vaiarelli A, Cimadomo D, Colamaria S, Alviggi C, Trabucco E, Venturella R, Vajta G, Rienzi L. Follicular versus luteal phase ovarian stimulation during the same menstrual cycle (DuoStim) in a reduced ovarian reserve population results in a similar euploid blastocyst formation rate: new insight in ovarian reserve exploitation. Fertil Steril. 2016 Jun;105(6):1488-1495.e1. doi: 10.1016/j.fertnstert.2016.03.002. Epub 2016 Mar 25. PMID 27020168